CLINICAL TRIAL: NCT02892305
Title: Hepatic Resection for Metastatic Pancreatic Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00073208
Record Dates: First submitted 2016-08-29; First posted 2016-09-08 (Estimated); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Pancreatic Neoplasms; Neoplasm Metastasis; Liver Metastases
Keywords: Pancreaticoduodenectomy; Hepatectomy; Liver ablation; Whipple
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis | interventions — Pancreaticoduodenectomy; Hepatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PAC with LVLM: Patients with pancreatic cancer and low-volume liver metastasis
  Interventions: Procedure: Hepatic Resection or Ablation with Pancreaticoduodenectomy

INTERVENTIONS:
Procedure: Hepatic Resection or Ablation with Pancreaticoduodenectomy — Patients will undergo pancreaticoduodenectomy, or the Whipple procedure, which involves removal of the head of the pancreas, the duodenum, and a portion of the stomach, as well as the gallbladder and a portion of the bile duct.
  The patient will also undergo a Hepatectomy, the surgical resection or removal of all or part of the liver or Microwave Ablation (MWA) if determined by the surgeon to be the best course of care.
  Other Names: Whipple; Hepatectomy; Microwave Ablation

SUMMARY:
The purpose of this study is to demonstrate the feasibility of an aggressive multimodal approach among patients with stage IV pancreatic cancer (PAC) with isolated, low-volume hepatic metastasis (LVHM). We will evaluate and describe the surgical and overall outcomes of an initial cohort of subjects who undergo pancreatectomy and hepatic resection/ablation for PAC with LVHM. The end of study results will be reviewed by the Hepatiobiliary Multidisciplinary Conference (HDMC) and Surgery Audit Committee (SAC) to determine the appropriateness of adding this treatment arm for patients with oligometastatic metastatic pancreatic cancer.

DETAILED DESCRIPTION:
This is a small interventional pilot study that will be conducted as a single-site study at Duke University Health System (DUHS). All subjects with pancreatic cancer and low-volume liver metastases (< or = 3 lesions) who meet criteria for pancreatic and liver resection will be offered the opportunity to participate. Potential subjects will be referred by the Medical Oncology physicians at Duke if they feel like the patient would be suitable for this study. We anticipate enrolling 15 subjects to include 10 evaluable subjects in the analysis.

Any subject who consents to the study will proceed with primary resection, including pancreaticoduodenectomy or distal pancreatectomy, and liver resection/ablation of the metastases.

Screening will include a medical record review, standard of care CT scan/MRI, clinical evaluation including physical, vitals, height weight and routine blood tests.

Preoperative data such as sex, race, age at resection, ASA class, race, body mass index (BMI), pretreatment staging, CA 19-9 (missing in open PD), tumor size (cm), and neoadjuvant therapy (no; yes), time to initiation and completion will also be captured.

Perioperative data like date of surgery, OR time, ASA class, intra-operative transfusion requirements, fluid administration, EBL, operative complications (including but not limited to infection, bleeding, need for re-operation, thrombus, pancreatic leak, bile leak, liver failure, nutritional data like use of TPN and tube feedings, and length of stay will be collected.

Post-operative data regarding re-admission and surveillance data for oncologic outcomes such as re-operation, final pathology margin status, nodal status, and postoperative CA 19-9, as well as DFS and OS, including date of death if applicable, during the provided follow up period.

To ensure accurate and complete incorporation of medical data, a database of perioperative outcomes will be prospectively maintained during the subject's hospital stay and for the first 3 months following surgery. Duke University is a member of the National Surgical Quality Improvement Program (NSQIP), with 100% participation in Hepatopancreaticobiliary (HPB) procedures. As such, all preoperative data and 30-day outcomes are collected by a fully trained Surgical Clinical Reviewer and are available within our electronic medical record (EMR). NSQIP provides a robust, audited dataset that has been validated to optimize the accuracy of data collection, substantially reducing the cost and resource requirements of data extraction. Following this 30-day period, data will be collected at regularly scheduled clinic visits, which typically occur weekly until 6-12 weeks post-surgery, then 3-4 months for the first year, and every 6 months thereafter and stored in a local, REDCap database.

Subjects' medical records will be continually reviewed for surgical complications and for overall survival (date of subject death).

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 18 years of age and at least the minimum Age of Majority according to applicable State or Country Law
* Subject is a surgical candidate, (i.e., is able to undergo general anesthesia and surgical resection for diagnosis of cancer)
* The Hepatobiliary Multidisciplinary Committee (HDMC) must approved of this intervention.
* Insurance pre-authorization must be received unless the subject decides to pay out of pocket..
* Subject has been informed of the study procedures and the treatment and has signed an informed consent form
* less than or equal to 3 liver lesions

Exclusion Criteria:

* Subject is not a suitable candidate for surgical intervention
* The Hepatobiliary Multidisciplinary Committee (HDMC) disapproves of this intervention.
* Insurance will not cover the procedure or subject not willing to pay out of pocket.
* Pregnant women
* Non-English speaking Subjects

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with biopsy-proven, or radiographically evident, resectable pancreatic head cancer who are found to have low-volume hepatic metastases at time of pancreaticoduodenectomy.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2018-05-18 (Actual); Primary Completion 2023-05-17 (Actual); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
90-day mortality | 90 days postoperatively
  Number of deaths within 90 days of operation
Disease Progression | up to 1 year postoperatively
  Time to disease progression
Overall Survival | up to 1 year postoperatively
  Number of months until death

SECONDARY OUTCOMES:
Postoperative length of stay | 90 days postoperatively
  Number of days in the hospital post-surgery
Frequency of pancreatic leak | 1-2 weeks postoperatively
  Number of leaks (Types A, B, C and bile)
Readmission to hospital | 90 days postoperatively
  Number of patients readmitted to the hospital post-operatively
Margin status | 90 days postoperatively
  Number of patients with positive margins
Lymph node status | 90 days postoperatively
  Number of positive lymph nodes
Time to Adjuvant therapy | Up to 5 years postoperatively
  Length of time to treatment after surgery
OR time | 1-2 days
  Length of time in the OR during surgery
Intraoperative estimated blood loss | 1-2 days
  Amount of blood loss during surgery in milliliters

CONTACTS AND LOCATIONS:
Overall Officials: Sabino Zani, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Argentiero A, Calabrese A, Sciacovelli AM, Delcuratolo S, Solimando AG, Brunetti O. Complete Response of Synchronous Liver Metastasis in a Pancreatic Ductal Adenocarcinoma, When Surgery Could Represent a Therapeutic Option. Can J Gastroenterol Hepatol. 2020 Oct 9;2020:8679751. doi: 10.1155/2020/8679751. eCollection 2020. PMID 33102398